CLINICAL TRIAL: NCT01476878
Title: Frameless Stereotactic Radiosurgery for Brain Metastases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alberta Health services (Other)
Collaborators: Tom Baker Cancer Centre (Other)
Responsible Party: Jon-Paul Voroney, Tom Baker Cancer Centre
Organization: AHS Cancer Control Alberta (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRAMELESS SRS
Record Dates: First submitted 2010-07-09; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-08

CONDITIONS: Brain Metastases
Keywords: Radiosurgery; Frameless radiosurgery; Accuracy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Arm (Experimental): Each study patient will receive high dose, single treatment radiation using a plastic mask instead of a head frame that pins into a patient's skull.
  Interventions: Device: Frameless Stereotactic Radiosurgery with radiation mask

INTERVENTIONS:
Device: Frameless Stereotactic Radiosurgery with radiation mask — Linac-based radiosurgery using a thermoplastic mask (single treatment)
  Other Names: Frameless Stereotactic Radiosurgery using radiation mask

SUMMARY:
The investigators plan to study high dose, single treatment radiation, using a plastic mask instead of a head frame that pins into a patient's skull. The investigators need to (1) quantify set-up accuracy and patient motion during radiation treatment and (2) ensure that without the head frame the tumour control rate and risk of complications are similar to our previous experience using the head frame.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain metastases from a biopsy-proven primary extra-cranial tumor site, excluding lymphoma, germ cell, and small cell lung carcinoma histologies.
* One to four metastases, and all lesions < 3.5 cm in maximal diameter. Extracranial metastases is of minimal volume or stable with treatment. - Karnofsky performance status ≥ 70

Exclusion Criteria:

* None of the lesions is abutting or within critical neurological structures: *brainstem

  * optic chiasm
  * eye, and optic nerve.
* The clearance between metastatic lesions and all critical structures must be at least 2 mm.
* Patients must not have leptomeningeal disease.
* Contraindications to imaging or radiation (e.g. pregnancy, elevated serum creatinine, allergy to contrast agents, severe claustrophobia, metal particles in the eye).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of patient movement occurring during treatment. | overall

SECONDARY OUTCOMES:
Local tumour control | overall
risk of complication (radionecrosis) | overall

CONTACTS AND LOCATIONS:
Overall Officials: Jon-Paul Voroney, MD, Principal Investigator — Tom Baker Cancer Centre
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada